CLINICAL TRIAL: NCT01191216
Title: A Phase 1 Study of 1-Methyl-D-tryptophan (NSC-721782) in Combination With Docetaxel in Metastatic Solid Tumors
Brief Title: 1-Methyl-D-Tryptophan and Docetaxel in Treating Patients With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02528; NCI-2011-02528 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000684389; MCC-16264; MCC16264 (Other: H. Lee Moffitt Cancer Center and Research Institute); 8784 (Other: CTEP); N01CM00100 (NIH); P30CA076292 (NIH)
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — 1-methyltryptophan; Docetaxel

ARMS (1):
- Arm I (Experimental): Patients receive oral 1-methyl-d-tryptophan twice daily on days 1-21 and docetaxel IV over 1 hour on day 1 (in course one patients receive 1-methyl-d-tryptophan once daily on days 1 and 3-21).
  Interventions: Drug: 1-methyl-d-tryptophan; Drug: docetaxel; Other: diagnostic laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: 1-methyl-d-tryptophan
  Other Names: indoximod
Drug: docetaxel
  Other Names: RP 56976; Taxotere; TXT
Other: diagnostic laboratory biomarker analysis
Other: pharmacological study
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of giving 1-methyl-d-tryptophan and docetaxel together in treating patients with metastatic solid tumors. Biological therapies, such as 1-methyl-d-tryptophan, may stop the growth of tumor cells by stimulating the immune system and by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving 1-methyl-d-tryptophan with chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The MTD of the 1-MT/docetaxel combination using CTCAE 4.0 criteria.

SECONDARY OBJECTIVES:

I. Determination of PK data for the combination of docetaxel plus oral 1-MT.Overall objective response rate (CR, PR) per RECIST criteria.

OUTLINE: This is a dose-escalation study.

Patients receive oral 1-methyl-d-tryptophan twice daily on days 1-21 and docetaxel IV over 1 hour on day 1 (in course one patients receive 1-methyl-d-tryptophan once daily on days 1 and 3-21). Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for pharmacokinetic and correlative studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic solid malignancy

  * Preference will be given to patients whose malignancies are treated with docetaxel as part of routine therapy
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan
* Patients with known brain metastases will only be eligible after their tumors have been treated with definitive resection and/or radiotherapy and they are neurologically stable for at least 1 month off steroids
* ECOG performance status ≤ 2 (Karnofsky ≥ 60%)
* Life expectancy of greater than 4 months
* Leukocytes ≥ 3,000/μL
* Absolute neutrophil count ≥ 1,500/μL
* Platelets ≥ 100,000/μL
* Total bilirubin normal
* AST/ALT ≤ 1.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Negative pregnancy test
* Not pregnant or nursing
* Sexually active women of child-bearing potential must agree to use two forms of contraception (hormonal and barrier method of birth control or abstinence) prior to study entry, for the duration of study participation, and for a minimum of 1 month after completion of the study; men should be discouraged from fathering children while on treatment
* No history of gastrointestinal disease causing malabsorption or obstruction such as, but not limited to, Crohn's disease, celiac sprue, tropical sprue, bacterial overgrowth/blind loop syndrome, gastric bypass surgery, strictures, adhesions, achalasia, bowel obstruction, or extensive small bowel resection
* No patients with any active autoimmune disease (i.e., psoriasis, extensive atopic dermatitis, asthma, IBD, M.S., uveitis, vasculitis), chronic inflammatory condition, or any condition requiring concurrent use of any systemic immunosuppressants or steroids for any reason

  * Mild-intermittent asthma requiring ONLY occasional beta-agonist inhaler use or mild localized eczema allowed
* No uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction or percutaneous coronary interventions within the last 6 months, cardiac arrhythmia, active autoimmune diseases, or major psychiatric illness/social situations that would limit compliance with study requirements as judged by the primary investigator at each site

  * Patients with well-controlled, chronic medical conditions under the supervision of the patient's primary physician (i.e., hypertension, hyperlipidemia, coronary heart disease, diabetes mellitus) are eligible
* No HIV-positive patients or those with other acquired/inherited immunodeficiencies
* No patients with more than one active malignancy at the time of enrollment
* No history of allergic reactions (significant urticaria, angioedema, anaphylaxis) attributed to compounds of similar chemical or biologic composition to 1-methyl-d-tryptophan (this wouldi nclude L-tryptophan or 5-hydroxy-tryptophan supplements) or history of severe hypersensitivity reactions to docetaxel or to other drugs formulated with polysorbate 80
* No patients with an allo-transplant of any kind (this would include those with a xenograft heart valve)
* No prior treatment with experimental systemic immunotherapies such as CTLA-4 mAb (with the exception of vaccines)
* No patients who have received any prior experimental active immunotherapy consisting of targeted monoclonal antibodies or pharmaceutical compounds

  * Patients who have received prior experimental vaccine may be enrolled if approved by the PI
  * Patients who have received commercially available active immunotherapies such as adjuvant interferon must have completed therapy over 1 year prior to enrollment and have no evidence of autoimmune sequelae
  * Prior therapy with approved monoclonal antibodies such as bevacizumab, cetuximab, panitumumab, or trastuzumab allowed
* No patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not have received docetaxel in the metastatic setting previously, but are eligible for the trial if they received docetaxel in the adjuvant setting and at least one year elapsed between completion of adjuvant chemotherapy and disease recurrence
* Patients may have received any number of prior chemotherapy treatments
* Patients may not be concomitantly receiving any other investigational agents or standard therapies with the intent of treating their malignancy while on study
* No supplements containing L-tryptophan or derivatives there of are allowed to be taken while on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose level in which 1 of 6 patients experiences DLT assessed using CTCAE version 4.0 | 21 days

SECONDARY OUTCOMES:
PK data | 0, 1, 2, 4, 8, 12, 24, and 48 hours
Overall objective response rate per RECIST criteria | From the start of the treatment until disease progression/recurrence
  The analysis will be descriptive in nature as it will include patients with metastatic solid tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Soliman, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (5):
- United States (5):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Billings Clinic, Billings, Montana
  - University of North Carolina, Chapel Hill, North Carolina
  - Virginia Commonwealth University, Richmond, Virginia